CLINICAL TRIAL: NCT02101983
Title: Feasibility of Outpatient Daily High Dose Cytarabine as Consolidation Therapy for Older Patients With Acute Myeloid Leukemia
Brief Title: Pilot Study of Feasibility of Outpatient Daily High Dose Cytarabine as Consolidation Therapy for Older Patients With Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Deborah Mulford, Associate Professor, University of Rochester
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 35606
Record Dates: First submitted 2013-10-14; First posted 2014-04-02 (Estimated); Results first posted 2018-06-27 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute myeloid leukemia; outpatient consolidation treatment
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Outpatient HiDAC Consolidation (Experimental): Patients will receive 2 cycles of 1.5 grams/m2/day of intravenous cytarabine once daily for six consecutive days. Toxicity will be monitored through the duration of treatment. Observation will be complete upon count recovery and resolution of toxicity after the second cycle.
  Interventions: Drug: Cytosine Arabinoside
- Quality of Life Comparison Group (Active Comparator): Patients receiving outpatient intravenous cytarabine will complete the EORTC QLQ-C30 quality of life form on the last day of each cycle of chemotherapy.
  Interventions: Drug: Cytosine Arabinoside

INTERVENTIONS:
Drug: Cytosine Arabinoside
  Other Names: AraC; Cytosar U; Cytosine aribinoside; Arabinosylcytosine; Cytarabine sterile; 1-B-Arabinoe-furanosyl-cytosine

SUMMARY:
High-dose cytarabine (HiDAC) is considered a standard chemotherapy treatment for patients with acute myeloid leukemia. However, most patients receiving this therapy are required to be admitted to the hospital during their treatment course.

The purpose of this study is to compare the safety and cost of high-dose cytarabine treatment given in an in-patient setting versus an out-patient setting.

DETAILED DESCRIPTION:
The primary objective of this study is to:

• To determine the incidence of grade 3 to 5 non-hematologic toxicity of high-dose cytarabine (HiDAC) for AML consolidation administered in an outpatient setting.

The secondary objectives of this study are to:

* To determine cost effectiveness of outpatient HiDAC consolidation versus the standard of care inpatient HiDAC consolidation.
* Evaluate patient quality of life (QOL) with this outpatient regimen in comparison to that with the standard inpatient regimen.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Outpatient Administration of HiDAC

* Unequivocal diagnosis of AML (>20% blasts in the bone marrow based on the WHO classification), excluding M3 (acute promyelocytic leukemia).
* Documented complete remission (CR) following induction chemotherapy as defined as (18):
* Bone marrow with <5% blasts; absence of blasts with Auer rods
* Absolute neutrophil count >1000/mcL
* Platelets >100,000/mcL
* Independence of red cell transfusions
* Absence of extramedullary disease
* Age ≥ 55 years.
* Relapsed AML patients are eligible as long as they meet other inclusion and exclusion criteria.
* Good performance status of (ECOG 0-2), see appendix 15.3.
* Adequate renal and hepatic function (Cr ≤ 1.2, alkaline phosphatase <3.0 x upper limit of normal, total bilirubin <1.5 x upper limit of normal unless there is a history of Gilbert's disease).

Inclusion Criteria for Quality of Life Comparison Group

* All patients decline to participate as an out-patient or who are not eligible for participation in the out-patient portion of the study will be approached to participate in the QOL comparison.
* Age ≥ 18 years

Exclusion Criteria:

Exclusion Criteria for All Patients

* Active, uncontrolled viral, bacterial, or fungal infection.
* Documented CNS leukemia.
* If unable to do a reliable cerebellar examination for monitoring of neurotoxicity.
* History of prior autologous or allogeneic bone marrow/stem cell transplant.
* New York Heart Association class III/IV congestive heart failure, see appendix 15.4, or active ischemic heart disease.
* Pregnant or lactating women (women and men of childbearing age should use effective contraception).
* Concomitant active malignancy requiring treatment with cytotoxic chemotherapy or radiation therapy. (Ongoing hormonal therapy for the treatment of malignancy would not exclude patients from this trial.)
* Time period of greater than 10 weeks between initiation of induction chemotherapy and day 1 of the first cycle of consolidation chemotherapy.
* Patients seropositive for infection with Human Immunodeficiency Virus (HIV) are excluded due to potential for serious infectious complications associated with T-cell suppressive therapy in these patients.

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-05; Primary Completion 2014-12 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Mulford, M.D., Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Outpatient HiDAC Consolidation: Patients will receive 2 cycles of 1.5 grams/m2/day of intravenous cytarabine once daily for six consecutive days. Toxicity will be monitored through the duration of treatment. Observation will be complete upon count recovery and resolution of toxicity after the second cycle.
  Cytosine Arabinoside
- Quality of Life Comparison Group: Patients receiving outpatient intravenous cytarabine will complete the EORTC QLQ-C30 quality of life form on the last day of each cycle of chemotherapy.
  Cytosine Arabinoside
Period: Overall Study
Arm/Group | Outpatient HiDAC Consolidation | Quality of Life Comparison Group
Started | 5 | 6
Completed | 4 | 6
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Outpatient HiDAC Consolidation | Quality of Life Comparison Group | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 6 | 10
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grades 3 to 5 Non-hematologic Toxicity.
Description: To determine the incidence of number of grades 3 to 5 non-hematologic toxicity of high-dose cytarabine for AML consolidation administered in an outpatient setting.
Time Frame: 3 months
Population: Subjects with a documented unequivocal diagnosis of AML in complete remission, age >/= 55 years, with good performance status and adequate renal and hepatic function. Subjects who are eligible for standard of care inpatient HiDAC consolidation will be approached to participate in the Quality of Life comparison group.
Measure: Count of Participants; unit: Participants
Arm/Group | Outpatient HiDAC Consolidation | Quality of Life Comparison Group
Number analyzed (Participants) | 4 | 5
Participants | 4 | 5

2. Secondary Outcome: Number of Participants Who Successfully Completed the of Quality of Life Form
Description: Subjects receiving outpatient high dose cytarabine or inpatient high dose cytarabine will complete the European Organization for Research and Treatment of Cancer Quality of Life tool on the last day of each cycle of chemotherapy. It encompasses 5 functional scales, 3 symptom scales and a global health measure. Scores range from 0-100 with higher scores associated with improved quality of life.
Time Frame: 3 months
Population: Subjects must have an unequivocal diagnosis of AML in a documented complete remission, age >/= 55 years with a good performance status and adequate renal and hepatic function. Subjects who decline participation as an outpatient will be approached to participate in the quality of life comparison group.
Measure: Count of Participants; unit: Participants
Arm/Group | Outpatient HiDAC Consolidation | Quality of Life Comparison Group
Number analyzed (Participants) | 4 | 5
Participants | 4 | 5

3. Secondary Outcome: Mean Cost Savings
Time Frame: 3 months
Population: Data was not collected from the participants for this outcome measure.
Arm/Group | Outpatient HiDAC Consolidation | Quality of Life Comparison Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Outpatient HiDAC Consolidation | Quality of Life Comparison Group
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/6
Other Adverse Events (participants affected / at risk) | 3/4 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Outpatient HiDAC Consolidation (N=4) | Quality of Life Comparison Group (N=6)
neutropenia (Blood and lymphatic system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Outpatient HiDAC Consolidation (N=4) | Quality of Life Comparison Group (N=6)
facial flushing (Vascular disorders) | 1 | 0
increased creatinine (Musculoskeletal and connective tissue disorders) | 1 | 0
increased alanine aminotransferase (Hepatobiliary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes